CLINICAL TRIAL: NCT03833375
Title: Shared Decision Making to Improve Goals-of-Care Decisions for Families of Severe Acute Brain Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Yale University (Other); University of Florida (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susanne Muehlschlegel, Associate Professor of Neurocritical Care, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H00004724/H00015764; 5K23HD080971 (NIH)
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Traumatic Brain Injury; Ischemic Stroke; Intracerebral Hemorrhage
Keywords: TBI; stroke; ICH; AIS; decision aid; shared decision making; neurocritical care; SABI; surrogate
MeSH Terms: conditions — Brain Injuries, Traumatic; Ischemic Stroke; Cerebral Hemorrhage; Stroke | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Open-label, usual-care-controlled feasibility trial comparing decision aid intervention prior to the goals-of-care family meeting to standard of care (no intervention prior to family meeting).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (n=20) (No Intervention): Control: general information about TBI from Center for Disease Control (CDC)/about stroke/Intracerebral Hemorrhage (ICH) from American Heart/Stroke Association
- Decision Aid (n=20) (Experimental): Paper Decision aid (share decision making tool) with worksheet for surrogates
  Interventions: Other: Decision Aid

INTERVENTIONS:
Other: Decision Aid — Shared-decision making tool
  Arms: Decision Aid (n=20)

SUMMARY:
Severe acute brain injury (SABI), including large artery acute ischemic stroke, intracerebral hemorrhage, and severe traumatic brain injury continue to be the leading cause of death and disability in adults in the U.S. Due to concerns for a poor long-term quality of life, withdrawal of mechanical ventilation and supportive medical care with transition to comfort care is the most common cause of death in SABI, but occurs at a highly variable rate (for example in Traumatic Brain Injury (TBI) 45-89%). Decision aids (DAs) are shared decision-making tools which have been successfully implemented and validated for many other diseases to assist difficult decision making. The investigators have developed a pilot DA for goals-of-care decisions for surrogates of SABI patients. This was developed through qualitative research using semi-structured interviews in surrogate decision makers of TBI patients and physicians. The investigators now propose to pilot-test a DA for surrogates of SABI patients in a feasibility trial.

DETAILED DESCRIPTION:
Severe acute brain injury (SABI), including large artery acute ischemic stroke, intracerebral hemorrhage, and severe traumatic brain injury continue to be the leading cause of death and disability in adults in the U.S, accounting for more than 200,000 of the acute brain injury-related deaths in the U.S. annually. Patients with SABI are critically ill and most commonly require mechanical ventilation and supportive medical care with artificial nutrition to ensure survival. However, due to concerns for a poor long-term quality of life, withdrawal of mechanical ventilation and supportive medical care with transition to comfort care is by far the most common cause of death in SABI but occurs at a highly variable rate (for example in TBI 45-90%) at different trauma centers. Shared decision making is a collaborative process that enhances patients' and surrogates' understanding about prognosis, encourages them to actively weigh the risks and benefits of a treatment, and to match them to patient preferences, thereby decreasing decisional conflict and improving decision quality and health related outcomes. Decision aids (DAs) are shared decision-making tools which have been successfully implemented and validated for many other diseases to assist difficult decision making. No DA currently exists for goals-of-care decisions in SABI. Such a patient- and family-centered DA has the potential to improve decision-making for SABI patients by ensuring proxies receive consistent, evidence-based prognostication while also addressing patients' preferences and values. The investigators have developed a pilot DA for goals of care decisions by surrogates of SABI patients using qualitative research using semi-structured interviews in surrogate decision makers of TBI patients and physicians, followed by an iterative feedback process with feedback by surrogates, physicians, and other stakeholders (ICU nurses). The investigators now propose to pilot-test a DA for surrogates of SABI patients in a feasibility trial.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age; no upper age limit
* Documented health care proxy or legal next of kin of admitted SABI patient with traumatic brain injury, intracerebral hemorrhage or acute ischemic stroke.
* ≥3 days after insult ("stabilization period"); clinical team may ask study team to wait longer if clinically indicated
* SABI patient remains "critically ill" after 3 days defined as: either intubated and mechanically ventilated, or unable to swallow, needing feeding tube beyond hospital discharge (even if not intubated)
* Surrogate is physically present in ICU to receive decision aid and participate in planned family meeting in person (not over phone)

Exclusion Criteria:

* Devastating SABI near death
* Patient will be extubated and pass swallow evaluation (as deemed by clinical team)
* Surrogate is non-English speaking and no interpreter available to translate decision aid (no available validated, translated decision aid version)
* Surrogate is illiterate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-02-11 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Recruitment | From date of approaching surrogate decision maker for consent until the date of the first documented goals-of-care family meeting, assessed up to 1 month after admission.
  Consent rate
Participation | 1-36 hours after family meeting
  Proportion of participants who read decision aid and completed worksheet
Retention | 3 months
  Number of participants who complete follow-up

SECONDARY OUTCOMES:
Clinician-surrogate concordance scale score | Baseline and 1-36 hours after family meeting
  measures prognostic concordance between ICU clinicians and surrogates. Participants from both groups will independently estimate numerically a SABI patient's 6-month survival and return to independence. Concordance is calculated as the absolute value of the difference in prognosis between the surrogate and the clinician, and, therefore, can range from 0 (no concordance) to 100 (full concordance).
Decision Self-Efficacy Scale | 1-36 hours after family meeting
  is a validated scale that measures self-confidence in making an informed choice using a 5-point Likert scale ranging from 0 (not at all confident) to 4 (very confident).
Decisional Conflict Scale | 1-36 hours after family meeting
  is a validated scale that measures the personal perception of choosing an option and factors contributing to choice uncertainty. It is a 16-item, 5-item Likert scale with sub-scores for uncertainty, feeling informed, values clarity, decision support and effective decision-making. It ranges from 0 (strongly agree) to 4 (strongly disagree).
AIS/Intracerebral Hemorrhage (ICH)/Traumatic Brain Injury (TBI) knowledge test | Baseline and 1-36 hours after family meeting
  Medical knowledge about the goals-of-care decision in SABI will be assessed using the medical knowledge test, which was adapted to 17 questions about goals-of-care and SABI, all of which are addressed in the decision aid. The % correct will be calculated.
Hospital Anxiety and Depression Scale (HADS) | Baseline,1-36 hours after family meeting, and 3-months
  is a 14-item, two-domain (depression, anxiety) instrument with reliability and validity among ICU surrogates, which is recommended by consensus guidelines for the prospective measurement of psychological distress among ICU surrogates. Each of the 14 questions are scored between 0 (not at all) and 3 (most of the time), and summed up for a total HADS score, which ranges from 0 to 42, with higher scores indicating worse symptoms. Total HADS 0-7 =normal, 8-10 borderline abnormal, 11-21=abnormal, indicating high anxiety and depression.
Impact of Events Scale-revised | Baseline,1-36 hours after family meeting, and 3-months
  is a is a validated 15-item instrument, measuring post-traumatic stress disorder (PTSD) symptoms. Total score is the sum of all questions and ranges from 0 to 88, with higher scores indicating worse PTSD symptoms.
Quality of Communications Scale | 1-36 hours after family meeting
  is a is a validated 17-item patient-centered instrument widely used in the ICU to assess surrogates' satisfaction of clinician communication about treatments and understanding treatment decisions. It ranges between 0 (poor) to 10 (absolutely perfect). Total score is the sum of all questions and ranges from 0 to 100, with higher scores indicating better communication.
Patient-Perceived Centeredness of Care Scale | 1-36 hours after family meeting
  is a is a validated 14-item, 4-point Likert scale based test. Its version adapted to surrogates has shown responsiveness in a recent trial of a nurse-driven communication intervention for surrogates in the ICU. It ranges between 1 (very well) to 4 (not at all), and median score is calculated from all questions. Median scores range from 1 to 4, with lower scores indicating more patient- and family-centered care.
Cumulative duration of the goals-of-care family meetings | 1-36 hours after family meeting
  Investigators will track the duration of each goals-of-care meeting. At the patient's ICU discharge, investigators will sum up the cumulative duration of all goals-of-care meetings [minutes].
Total number of goals-of-care family meetings | 1-36 hours after family meeting
  Investigators will sum up the total number of goals-of-care meetings at the patient's ICU discharge.
Patient's survival status | 3-months after goals of care decision
  Investigators will record whether the patient is dead or alive.
Patient's Glasgow Outcome Scale | 3-months after goals of care decision
  The Glasgow Outcome Score (GOS) is a validated 5-point scale given to traumatic brain injury or other brain injury patients at some point in their recovery. It is a very general assessment of the general functioning of the person who suffered a head injury or other neurological injury. It ranges from 1-5 (higher scores indicating better functional status): 1=death, 2=Vegetative State, 3=Severely Disabled (conscious but the patient requires others for daily support due to disability), 4=Moderately Disabled (the patient is independent but disabled), 5=Good Recovery (the patient has resumed most normal activities but may have minor residual problems).
Patient's modified Rankin Scale | 3-months after goals of care decision
  is a validated scale that measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It ranges from 0 (no symptoms at all) to 6 (death).
Surrogate Decision Regret Scale | 3-months after goals of care decision
  is a validated scale that measures distress or remorse after a health care decision with high internal consistency. It asks 5 questions and provides a 5-point Likert scale. It ranges between 1 (strongly agree) to 5 (strongly disagree).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Susanne Muehlschlegel, MD, MPH, Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - Yale Medical School/Yale New Haven Medical Center, New Haven, Connecticut
  - University of Massachusetts Medical School, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quinn T, Moskowitz J, Khan MW, Shutter L, Goldberg R, Col N, Mazor KM, Muehlschlegel S. What Families Need and Physicians Deliver: Contrasting Communication Preferences Between Surrogate Decision-Makers and Physicians During Outcome Prognostication in Critically Ill TBI Patients. Neurocrit Care. 2017 Oct;27(2):154-162. doi: 10.1007/s12028-017-0427-2. PMID 28685395
- [Background] Moskowitz J, Quinn T, Khan MW, Shutter L, Goldberg R, Col N, Mazor KM, Muehlschlegel S. Should We Use the IMPACT-Model for the Outcome Prognostication of TBI Patients? A Qualitative Study Assessing Physicians' Perceptions. MDM Policy Pract. 2018 Mar 26;3(1):2381468318757987. doi: 10.1177/2381468318757987. eCollection 2018 Jan-Jun. PMID 30288437
- [Background] Muehlschlegel S, Shutter L, Col N, Goldberg R. Decision Aids and Shared Decision-Making in Neurocritical Care: An Unmet Need in Our NeuroICUs. Neurocrit Care. 2015 Aug;23(1):127-30. doi: 10.1007/s12028-014-0097-2. PMID 25561435
- [Background] Cai X, Robinson J, Muehlschlegel S, White DB, Holloway RG, Sheth KN, Fraenkel L, Hwang DY. Patient Preferences and Surrogate Decision Making in Neuroscience Intensive Care Units. Neurocrit Care. 2015 Aug;23(1):131-41. doi: 10.1007/s12028-015-0149-2. PMID 25990137
- [Derived] Muehlschlegel S, Goostrey K, Flahive J, Zhang Q, Pach JJ, Hwang DY. Pilot Randomized Clinical Trial of a Goals-of-Care Decision Aid for Surrogates of Patients With Severe Acute Brain Injury. Neurology. 2022 Oct 3;99(14):e1446-e1455. doi: 10.1212/WNL.0000000000200937. PMID 35853748